CLINICAL TRIAL: NCT01431742
Title: An Open Label, Longterm Treatment Evaluation of the Safety and Efficacy of BEMA® Buprenorphine in Subjects With Moderate to Severe Chronic Low Back Pain
Brief Title: Longterm Safety Study of BEMA Buprenorphine in Subjects With Chronic Low Back Pain
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: BioDelivery Sciences International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUP-306
Record Dates: First submitted 2011-09-08; First posted 2011-09-12 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Pain; Low Back Pain
Keywords: buccal soluble film; Pain; Back Pain; Low Back Pain; Buprenorphine; Analgesics, Opioid; Analgesics
MeSH Terms: conditions — Pain; Low Back Pain; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BEMA Buprenorphine (Experimental): buprenorphine buccal soluble film
  Interventions: Drug: BEMA Buprenorphine

INTERVENTIONS:
Drug: BEMA Buprenorphine — buccal soluble film; applied to the buccal mucosa twice daily
  Other Names: buprenorphine buccal soluble film

SUMMARY:
This is an open label study of up to approximately 52 weeks duration to assess the safety and effectiveness of BEMA Buprenorphine in the management of moderate to severe chronic low back pain.

BEMA Buprenorphine is an oral transmucosal form of the opioid analgesic, buprenorphine hydrochloride, intended for application to the buccal mucosa. Buprenorphine is a synthetic opioid that is classified as a partial μ-receptor agonist and a Schedule III controlled substance in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant and non-nursing female aged 18 or older
* History of moderate to severe chronic low back pain for ≥3 months with a pain intensity ≥5 [11 point NRS] reported during screening following discontinuation of current pain medication (opioids and NSAIDs) AND currently taking ≥10 mg oral morphine equivalent/day for ≥2 weeks
* Stable health, as determined by the Investigator, on the basis of medical history, physical examination, and laboratory results so as to comply with all study procedures
* Female subjects of childbearing potential must be using a recognized effective method of birth control
* Written informed consent obtained prior to any procedure being performed

Exclusion Criteria:

* Cancer related pain
* Reflex sympathetic dystrophy or causalgia (complex regional pain syndrome), acute spinal cord compression, cauda equina compression, acute nerve root compression, meningitis, or discitis
* Surgical procedure for pain within 2 months, or nerve/plexus block within 4 weeks, prior to titration period Day 0/1 visit
* History of severe emesis with opioids
* Clinically significant sleep apnea in the judgment of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Mean change in pain intensity | Baseline up to approximately Week 52
  The average of the visit pain scores for Baseline up to approximately Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Finn, PharmD, Study Chair — BioDelivery Sciences International
Locations (1):
- Marietta, Georgia, United States